CLINICAL TRIAL: NCT01125085
Title: A Prospective Non-randomized Study of 131I-L19SIP Radioimmunotherapy (RIT) in Combination With Whole Brain Radiation Therapy (WBRT) in Patients With Multiple Brain Metastases From Solid Tumors
Brief Title: 131I-L19SIP Radioimmunotherapy (RIT) in Combination With External Beam Radiation in Patients With Multiple Brain Metastases From Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19SIPI131-01/09; 2009-013002-13 (EudraCT Number)
Record Dates: First submitted 2010-05-12; First posted 2010-05-18 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Brain Metastases From Solid Tumors
Keywords: I131; L19; antibody; monoclonal; multiple brain metastasis; tumor targeting; radioimmunotherapy; Patients with brain metastases of solid tumors (>1), who are not amenable for surgical excision or stereotactic radiosurgery.
MeSH Terms: interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131I-L19SIP RIT in Combination with WBRT (Other): 131I-L19SIP Radioimmunotherapy (RIT) in Combination With Whole Brain Radiation Therapy (WBRT)
  Interventions: Radiation: 131I-L19SIP Radioimmunotherapy (RIT) in Combination With Whole Brain Radiation Therapy (WBRT)

INTERVENTIONS:
Radiation: 131I-L19SIP Radioimmunotherapy (RIT) in Combination With Whole Brain Radiation Therapy (WBRT) — * Patients will be treated with WBRT administering a total dosage of 30 Gy in fractions of 3 Gy
  * Dosimetric evaluation with 131I-L19SIP or 124I-L19SIP will be performed to assess eligibility for RIT.
  * Patients eligible for RIT will receive a therapeutic dose of 131I-L19SIP.
  * Total treatment duration is up to 4 weeks

SUMMARY:
The aim of this Proof of Concept study is to determine the therapeutic potential of the L19SIP antibody, labeled with the radionuclide 131I in combination with external beam radiation, for the treatment of patients with multiple brain metastases following the promising results with this agent in previous clinical studies.

The L19SIP antibody is a fully human antibody, capable of preferential localization around tumor blood vessels while sparing normal tissues. The formation of new blood vessels is a rare event in the adult (exception made for the female reproductive cycle), but is a pathological feature in most aggressive types of cancer. The presented study follows a Phase I and a subsequent Phase I/II dose finding and efficacy study with the same agent in patients with a variety of cancers where 131I-L19SIP had shown an excellent tolerability and therapeutic benefit for some patients enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* 6.3.1 Inclusion Criteria for Dosimetric Study Part (diagnostic 131I-L19SIP or 124I-L19SIP) and therapeutic study part
* Unresectable multiple brain metastasis from histologically or cytologically confirmed solid tumors. In exceptional cases also patients with a single brain metastasis if not amenable for surgical treatment might be included.
* Males or females, age > 18 years
* Measurable disease defined as at least one metastatic brain lesion that can be accurately and serially measured by the modified RECIST criteria (version 1.1)
* Prior therapy for metastatic disease allowed
* RPA Class II
* Life expectancy of at least 12 weeks
* Serum creatinine < 1.5 x ULN
* All toxic effects of prior therapy must have resolved to ≤ Grade 1 unless otherwise specified above
* Negative serum pregnancy test (for women of child-bearing potential only) at screening
* If of childbearing potential, agreement to use highly effective contraceptive methods (e.g., established use of oral, injected or implanted hormonal methods, placement of intrauterine device or intrauterine system, use of condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization or true abstinence) beginning at the screening visit and continuing until 3 months following last treatment with study drug.
* In case of treated males (including men who have had vasectomies) who have a partner who is pregnant or of child-bearing potential, agreement to use condoms beginning at the screening visit and continuing until 3 months following last treatment with study drug.
* Patients with microhaemorrhage can be included if the microhaemorrhage does not appear to significantly contribute to symptoms caused by the particular brain lesion and if the microhaemorrhage does not appear to significantly contribute to a possible mass effect of the brain lesion in question.

Additional Inclusion Criteria for Therapeutic Study Part

* Absolute neutrophil count > 1.0 x 109/L, hemoglobin > 8.0 g/dL (packed red cell transfusions allowed), and platelets > 100 x 109/L
* Total bilirubin ≤ 30 µmol/L (or ≤ 2.0 mg/dL). For patients with liver involvement with tumor total bilirubin ≤ 45 µmol/L (or ≤ 3.0 mg/dL).
* ALT and AST ≤ 2.5 x the upper limit of normal (10 x ULN for patients with hepatic involvement with tumor

Exclusion Criteria:

* Primary ocular melanoma
* Patients with brain metastasis amenable for surgical excision or stereotactic irradiation (radiosurgery)
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (TA, Tis & Ti) or any cancer curatively treated < 5 years prior to study entry
* Patients with history of whole brain irradiation
* History of HIV infection or infectious hepatitis B or C
* Presence of active infections (e.g. requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or interfere with the study.
* Inadequately controlled cardiac arrhythmias including atrial fibrillation
* Heart insufficiency (> Grade II, New York Heart Association (NYHA) criteria)
* Uncontrolled hypertension
* Ischemic peripheral vascular disease (Grade IIb-IV)
* Severe diabetic retinopathy
* Active autoimmune disease
* History of organ allograft or stem cell transplantation
* Recovery from major trauma including surgery within 4 weeks prior to administration of study treatment
* Pregnant woman
* Breast feeding female
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment
* Growth factors or immunomodulatory agents within 7 days of the administration of study treatment
* Patients in need of systemic treatment associated with a moderate or significant potential of hematotoxicity for rapidly progressive systemic disease during study treatment and up to 4 weeks after injection of therapeutic 131I-L19SIP.
* Hyperthyroidism or autonomous thyroid nodule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Uptake of 131I-L19SIP or 124I-L19SIP | 2 days
  Selective uptake of 131I-L19SIP or 124I-L19SIP in brain lesions
Safety of combined administration of 131I-L19SIP and whole brain radiation therapy (WBRT) | 13 months
  Safety will be assessed through physical examinations, vital signs, laboratory tests (including serum chemistries, hematology parameters) and the recording of adverse events. Treatment emergent adverse events will be summarized by CTCAE version 3 (and if possible by the RTOG/EORTG scale) and worse grade for all treated patients. Laboratory values and change in vital signs will be summarized.

SECONDARY OUTCOMES:
Overall response | 12 months
  Intracranial, extra cranial and overall response
Overall survival | 12 months
Clinical performance index in terms of Graded Prognostic Assessment (GPA) | 12 months
  GPA score will be assessed at the screening visit, during treatment and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Secondo Lastoria, Dr, Principal Investigator — ISTITUTO NAZIONALE PER LO STUDIO E LA CURA DEI TUMORI FONDAZIONE GIOVANNI PASCALE DI NAPOLI; Paul Mullholand, Dr, Principal Investigator — UCLH, Department of Cancer Medicine, London (UK)
Locations (10):
- Italy (8):
  - Irccs Centro Di Riferimento Oncologico (Cro) - Aviano, Aviano
  - Ospedali Riuniti Di Bergamo, Bergamo
  - Azienda Ospedaliero UNIVERSITARIA CAREGGI DI FIRENZE, Florence
  - ASUR Zona Territoriale 9, Medicina Nucleare Ospedale di Macerata, Macerata
  - Istituto Nazionale Per Lo Studio E La Cura Dei Tumori Fondazione Giovanni Pascale Di Napoli, Napoli
  - Arcispedale Santa Maria Nuova Di Reggio Emilia, Reggio Emilia
  - Irccs Istituto Clinico Humanitas, Rozzano (mi)
  - Irccs Ospedale Casa Sollievo Della Sofferenza - San Giovanni Rotondo, San Giovanni Rotondo (FG)
- United Kingdom (2):
  - Barts and the London NHS Trust Hospital, London
  - UCLH, Department of Cancer Medicine, London, London

REFERENCES:
- [Derived] Poli GL, Bianchi C, Virotta G, Bettini A, Moretti R, Trachsel E, Elia G, Giovannoni L, Neri D, Bruno A. Radretumab radioimmunotherapy in patients with brain metastasis: a 124I-L19SIP dosimetric PET study. Cancer Immunol Res. 2013 Aug;1(2):134-43. doi: 10.1158/2326-6066.CIR-13-0007. Epub 2013 May 20. PMID 24777501